## Impact of Liraglutide 3.0 on Body Fat Distribution—Statistical Analysis Plan

NCT 03038620

July 28, 2020

## Statistical Analysis Plan - Impact of Liraglutide 3.0 on Body Fat Distribution

#### Important points:

- 1. Modified intention-to-treat (mITT) which includes data from the full-analysis set of all participants who underwent randomization and had a follow-up endpoint assessment (full analysis set, FAS).
- 2. Secondary analyses will be performed using per-protocol approach which includes data from the full-analysis set of all participants who underwent randomization, received at least one dose of study drug, <u>and</u> completed a final imaging visit at the planned study end; this is termed a "completers analysis".
- 3. Missing values will be imputed with the Monte Carlo Markov Chain method. Sensitivity analyses will be performed to determine the effect of missingness/imputation on the primary and secondary outcomes.

## Descriptive:

- 1. Baseline characteristics of study population overall and stratified by treatment assignment
- 2. Mean medication adherence as a percentage of drug taken/drug dispensed after randomization through final outcomes assessment.
- 3. Proportion losing  $\geq$  5% body weight and  $\geq$  10% body weight in each group (and compared with p-value).
- 4. Adverse events: a) most frequent (%), b) serious (%), rate of withdrawal in each group for adverse events

#### Endpoints analysis:

Note: All to be reported as mean  $\pm$  standard deviation in each group with between group differences reported as placebo-adjusted difference with 95% confidence interval.

1. Primary endpoint: Relative percent change in visceral adipose tissue volume

## 2. Secondary endpoints

- a. Absolute change in visceral adipose tissue volume
- b. Relative percent change in body weight
- c. Absolute change in body weight
- d. Relative percent change in waist circumference
- e. Absolute change in waist circumference
- f. Relative percent change in total body adipose tissue volume
- g. Absolute change in total body adipose tissue volume
- h. Relative percent change in abdominal subcutaneous adipose tissue volume
- i. Absolute change in abdominal subcutaneous adipose tissue volume

- j. Relative percent change in lower body subcutaneous adipose tissue volume
- k. Absolute change in lower body subcutaneous adipose tissue volume
- 1. Relative percent change in liver fat percent
- m. Absolute change in liver fat percent
- n. Relative percent change in total body lean volume
- o. Absolute change in total body lean volume
- p. Relative percent change in total thigh muscle volume
- q. Absolute change in total thigh muscle volume
- r. Relative percent change in mean anterior thigh muscle fat infiltration percent
- s. Absolute change in mean anterior thigh muscle fat infiltration percent

### 3. Subgroup analyses

- a. To be performed for the primary endpoint as well as selected secondary endpoints as below:
  - i. Relative percent change in abdominal subcutaneous adipose tissue volume
  - ii. Relative percent change in lower body subcutaneous adipose tissue volume
  - iii. Relative percent change in liver fat percent
  - iv. Relative percent change in total thigh muscle volume
  - v. Relative percent change in mean anterior thigh muscle fat infiltration percent
- b. Age (stratified by median)
- c. Sex (M/F)
- d. Race (non-Hispanic black, non-Hispanic white, Hispanic)
- e. Body mass index (kg/m²) category (overweight 25-29.9, class I 30-34.9, class II/III ≥35)
- f. Sex-specific tertiles of total body fat (T1, T2, T3)
- g. Prediabetes (Y/N)

# 4. Correlation between change in body weight, BMI, total body fat, and change in fat distribution for:

- a. Visceral adipose tissue
- b. Abdominal subcutaneous adipose tissue
- c. Lower body subcutaneous adipose tissue
- d. Liver fat
- e. Anterior thigh muscle fat infiltration

#### 5. "Responders" analysis

- a. Pre-specified analysis stratified by those who did vs. did not lose ≥4% body weight at week 16 of treatment to determine differential outcomes among "responders" vs. "non-responders" as outlined in the Liraglutide package insert.
- b. This analysis will be performed for the primary endpoint only.

#### **Statistical approach:**

1. For continuous endpoints, an analysis of covariance model will be used to analyze mean changes. The model will include treatment, sex, BMI stratification ( $<30, \ge 30$ ),

- prediabetes status at baseline, interaction between BMI and prediabetes status strata as fixed effects, with the baseline value of the relevant variable as a covariate.
- 2. For categorical endpoints, logistic regression will be used with the same fixed effects and covariates as the analysis of covariance model.
- 3. Sensitivity analyses for primary endpoint

| Endpoint | Type of analysis | Description |
|---|---|---|
| Relative percent change in | mITT | Analysis of FAS with a valid |
| visceral adipose tissue | | non-imputed measurement at |
| | | study end |
| Relative percent change in | LOCF | Same analysis as the primary |
| visceral adipose tissue | | applied to all randomized |
| | | patients allowing for baseline |
| | | carried forward for those |
| | | without a post-baseline |
| | | measurement |
| Relative percent change in | MCMC | Same analysis as the primary |
| visceral adipose tissue | | applied to all randomized |
| | | patients allowing for |
| | | imputation of missing |
| | | observations using a |
| | | modeling method |

FAS denotes full analysis set, defined as all participants who underwent randomization and had a follow-up endpoint assessment